CLINICAL TRIAL: NCT02707770
Title: The Role of Ambulatory Oxygen in Improving the Effectiveness of Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Diseases Patients
Brief Title: The Role of Ambulatory Oxygen in Improving the Effectiveness of Pulmonary Rehabilitation for COPD Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for the study finished before anticipated participants enrolled
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15SM3060
Record Dates: First submitted 2016-02-23; First posted 2016-03-14 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Chronic Obstructive Pulmonary Diseases
Keywords: COPD, pulmonary rehabilitation, ambulatory oxygen therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambulatory oxygen (Experimental): Patient will use ambulatory oxygen during pulmonary rehabilitation programme (flow rate determined at the initial assessment to a maximum flow rate of 6 litres per minute)
  Interventions: Other: Pulmonary Rehabilitation
- Room air (Placebo Comparator): Patient will breath on room air during pulmonary rehabilitation programme
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation

SUMMARY:
Pulmonary rehabilitation (PR) is an exercise program tailored for patients with chronic lung disease that is a core part of the management of patients with Chronic Obstructive Pulmonary Disease (COPD). Many COPD patients develop low oxygen levels (desaturation) during exercise and this is often discovered when they are being evaluated for PR. Current practice is to administer oxygen to COPD patients with exercise-induced desaturation, but this is based on very limited evidence. This limited evidence relates to a short-term increase in exercise capacity and it is not known if this translates into longer term increases in activity or whether providing these patients with oxygen improves outcomes after PR.

In addition it is not known if patients given ambulatory oxygen continue to use it after completing PR. Evidence for a beneficial effect of oxygen would provide a more solid evidence base for its use. Conversely demonstration of no effect would allow reassessment of the use of oxygen and whether the costs are justified. Therefore the aims of this study are to assess the effects of oxygen on outcomes from PR and assess the usage of ambulatory oxygen following completion of PR.

DETAILED DESCRIPTION:
The study will be a randomised, single-blinded study comparing oxygen with air in Chronic Obstructive Pulmonary Disease (COPD) patients undergoing Pulmonary Rehabilitation (PR).

The study subjects will be patients with a confirmed diagnosis of COPD who have been accepted for PR and who are not hypoxemic at rest, but have exercise-induced desaturation (defined as a fall in oxygen saturations (SaO2) ≥4% to at least <90%, or any fall to a SaO2 <90%) and demonstrate positive improvement with use of ambulatory oxygen as per the British Thoracic Society 2015 Oxygen guidelines. It is standard practice for patients to have this assessment prior to commencing PR and as part of the assessment the flow rate required to increase the SaO2 to ≥90% during exercise will be determined. Patients will be recruited from PR programs at imperial college health care trust hospitals.

The subjects will be randomised to receive either oxygen at the flow rate determined at the initial assessment to a maximum flow rate of 6 litres per minute, or room air. The subjects will then undergo a standard program of PR over 6 - 8 weeks and then undergo reassessment. 20 patients are required in each group to detect a 30% effect size on the 6 minute walk test (6MWT) with 80% power at the 5% significance level and 29 patients in each group to detect a 25% effect with 80% power. Therefore a minimum of 20 patients per group will be included.

Baseline assessments prior to commencing PR will include symptom and quality of life assessments including Borg scale for assessment of breathlessness, Chronic Respiratory Questionnaire (CRQ), COPD Assessment Tool (CAT) and the Hospital Anxiety and Depression score (HAD). A 6 minute walk test (6MWT) will be carried out as this is a widely used and well validated tool to measure exercise capacity. A handheld dynamometer will be used to obtain more detailed measures of quadriceps muscle strength. In addition we will measure activity at home during and after PR using pedometers as this has never been investigated previously.These are simple devices that can be attached to patients and count the numbers of steps during a day and therefore provide an estimate of activity in the home environment. A yamax Digi-walker SW-200 pedometer will be used to count the number of steps taken per day. Patients will be instructed to wear the device on left side of the body all the time, except when sleeping or showering. Pedometer placement was standardised by placing it on the belt or waistband, in the midline of the thigh, consistent with the manufacturers recommendation and with other studies conducted previously. Patients will be record daily step counts on daily diary cards until their final follow up.

The measures of exercise capacity at the follow up assessment will be carried out off oxygen and will be carried out by an observer blinded as to whether they received oxygen or not during PR. All patients will be provided with ambulatory oxygen for domiciliary use after completing PR.

The hypothesis is that use of oxygen in selected patients improves exercise capacity during PR. The measurable aims will be exercise capacity and on-going usage of oxygen in this patient group.

Primary Objective

Assess the effects of ambulatory oxygen on outcomes from Pulmonary Rehabilitation

Secondary Objectives

1. Assess the proportion of patients that wish to continue to use ambulatory oxygen.
2. Assess the usage of ambulatory oxygen following completion of Pulmonary Rehabilitation
3. Assess whether initiation of ambulatory oxygen before or after PR has any influence on adherence to usage at 8 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
2. Fulfil the clinical criteria for Pulmonary Rehabilitation (PR)
3. Demonstrate exercise-induced desaturation (defined as a fall in SaO2 ≥4% to at least <90%, or any fall to a SaO2 <90%) and demonstrate positive improvement with use of ambulatory oxygen as per the British Thoracic Society 2015 Oxygen Guidelines

Exclusion Criteria:

1. Use of long term oxygen therapy
2. Unable to provide informed consent
3. Significant respiratory disease other than COPD
4. Any patient needing more than 6 litres per minute oxygen to correct desaturation
5. Severe desaturation: SaO2 < 80% during 6 Minute Walk Test
6. Any absolute contraindication to Pulmonary Rehabilitation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijayaragavan Padmanaban, MPT, Principal Investigator — Imperial healthcare NHS Trust
Locations (1):
- St Marys Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Ambulatory Oxygen: Patient will use ambulatory oxygen during pulmonary rehabilitation programme (flow rate determined at the initial assessment to a maximum flow rate of 6 litres per minute)
  Pulmonary Rehabilitation
- Room Air: Patient will breath on room air during pulmonary rehabilitation programme
  Pulmonary Rehabilitation
Period: Overall Study
Arm/Group | Ambulatory Oxygen | Room Air
Started | 10 | 10
Completed | 9 (One patient withdrew from the study following consent, initial assessment and randomisation) | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambulatory Oxygen | Room Air | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Full Range); unit: years] | 73 [54 to 80] | 72 [60 to 90] | 72.5 [54 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 7 | 4 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Exercise Capacity
Description: 6 Minute Walk Test (6MWT)- Distance in meters
Time Frame: 0, 8weeks
Measure: Mean (Full Range); unit: meters
Arm/Group | Ambulatory Oxygen | Room Air
Number analyzed (Participants) | 9 | 10
meters
  Baseline -0 | 332 [170 to 430] | 335 [140 to 500]
  Post PR - 8weeks | 346 [200 to 430] | 340 [140 to 510]

2. Secondary Outcome: Number of Participants Reporting a Change in the Quality of Life
Description: Chronic Respiratory Questionnaire(CRQ)- Number of Participants achieving minimal clinically important difference (MCID) in CRQ compared between baseline and follow up assessment.
Time Frame: 0,8weeks
Measure: Number; unit: participants
Arm/Group | Ambulatory Oxygen | Room Air
Number analyzed (Participants) | 9 | 10
participants | 3 | 2

3. Secondary Outcome: Number of Participants Reporting a Change in Anxiety Score
Description: Hospital anxiety and depression score- Anxiety component (HADS-A)-Numbers of participants achieving Minimal clinically important difference in HADS-A compared between baseline and follow up assessment.
Time Frame: 0,8weeks
Measure: Number; unit: participants
Arm/Group | Ambulatory Oxygen | Room Air
Number analyzed (Participants) | 9 | 10
participants | 4 | 3

4. Secondary Outcome: Number of Participants Reporting Change in Depression Score
Description: Hospital anxiety and depression score- Depression component (HADS-D)-Numbers of participants achieving Minimal clinically important difference in HADS-D compared between baseline and follow up assessment.
Time Frame: 0,8weeks
Measure: Number; unit: participants
Arm/Group | Ambulatory Oxygen | Room Air
Number analyzed (Participants) | 9 | 10
participants | 2 | 2

5. Secondary Outcome: Number of Participants Reporting Change in Chronic Obstructive Pulmonary Diseases Assessment Test (CAT)
Description: Chronic Obstructive Pulmonary diseases Assessment Test (CAT score)-Numbers of participants achieving Minimal clinically important difference in CAT score compared between baseline and follow up assessment.
Time Frame: 0,8weeks
Measure: Number; unit: participants
Arm/Group | Ambulatory Oxygen | Room Air
Number analyzed (Participants) | 9 | 10
participants | 5 | 3

6. Secondary Outcome: Number of Patients Reporting Change in Physical Activity
Description: Pedometer- Number of step counts
Time Frame: 8 weeks
Population: Due to technical problems identified with accuracy of device, this outcome measure was excluded from study
Arm/Group | Ambulatory Oxygen | Room Air
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Change in Quadriceps Muscle Strength
Description: Handheld Muscle testing- Number of participants achieving Minimal clinical important difference in quadriceps muscle strength compared between baseline and follow up assessment
Time Frame: 0,8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Oxygen | Room Air
Number analyzed (Participants) | 8 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event monitored throughout the study period ( Up to end of final follow up, approximately 8 weeks)
Description: Definition of AE is not different to clinicaltrials.gov definitions
Arm/Group | Ambulatory Oxygen | Room Air
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

LIMITATIONS AND CAVEATS:
Due to study terminated prematurely, unable to recruit the intended number of participants and complete extra follow ups as proposed in the study protocol.

Due to technical issue with pedometer device and validity of measurements, physical activity measurement was not included or analysed as part of the secondary outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT02707770/Prot_SAP_000.pdf